CLINICAL TRIAL: NCT00004642
Title: Phase I/II Study of Human Anti-Cytomegalovirus (CMV) Monoclonal Antibody MSL-109 in Newborns With Symptomatic Congenital CMV Infection Without Central Nervous System Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11673; NIAID-3748
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-03

CONDITIONS: Cytomegalovirus Infections
Keywords: congenital cytomegalovirus infection; cytomegalovirus infection; herpesvirus infection; immunologic disorders and infectious disorders; neonatal disorders; rare disease; viral infection
MeSH Terms: conditions — Cytomegalovirus Infections; Herpesviridae Infections; Immune System Diseases; Communicable Diseases; Infant, Newborn, Diseases; Rare Diseases; Virus Diseases | interventions — sevirumab

INTERVENTIONS:
Drug: SDZ MSL-109

SUMMARY:
OBJECTIVES: I. Evaluate the safety, tolerance, and potential efficacy of 3 doses of human anti-cytomegalovirus (CMV) monoclonal antibody SDZ MSL-109 (MOAB MSL-109) in the treatment of newborns with congenital CMV infection and no central nervous system disease.

II. Determine the relationship between plasma concentrations of MOAB MSL-109 and therapeutic outcome.

III. Determine whether MOAB MSL-109 influences the antibody response and clearance of virus from the urine.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are treated with human anti-cytomegalovirus monoclonal antibody MSL-109, administered intravenously every other week for a total of 3 doses.

Groups of 6 patients are treated at each of 3 MSL-109 doses; there is no intrapatient escalation.

No concurrent therapy with antibiotics for systemic infection, parenteral antifungal agents, biological response modifiers, or other antiviral agents is allowed.

Patients are followed every 2 weeks for 6 weeks, every 4 weeks for 12 weeks, then annually for 5 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Symptomatic congenital cytomegalovirus (CMV) infection confirmed by urine culture No CMV acquired natally or postnatally Normal eye exam and skull x-ray, computerized tomography, or magnetic resonance imaging No evidence of central nervous system CMV, e.g.: Microcephaly, hydrocephaly, or hydranencephaly Intracranial calcification Chorioretinitis Normal cerebrospinal fluid Preterm: WBC no greater than 30 Protein less than 120 mg/dL Term: WBC no greater than 25 Protein less than 80 mg/dL --Prior/Concurrent Therapy-- At least 2 weeks since investigational drugs No prior or concurrent antiviral agents --Patient Characteristics-- Life expectancy: No imminent demise Renal: Creatinine no greater than 1.5 mg/dL Other: Birth weight at least 1200 g No congenital toxoplasmosis, congenital rubella, or syphilis No active systemic infection, i.e.: Bacterial Non-CMV viral, including HIV Protozoal Fungal No severe concurrent clinical condition, e.g.: Non-CMV congenital disease Genetic abnormality Moderate to severe hyaline membrane disease

Ages: 0 Years to 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1995-02

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Whitley, Study Chair